CLINICAL TRIAL: NCT00086346
Title: A Randomized, Open-Label, Comparative Evaluation of Conversion From Calcineurin Inhibitor Treatment to Sirolimus Treatment Versus Continued Calcineurin Inhibitor Treatment in Liver Allograft Recipients Undergoing Maintenance Therapy
Brief Title: Study Evaluating of Calcineurin Inhibitor and Sirolimus (Rapamune) Treatment in Liver Transplant Recipients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-313
Record Dates: First submitted 2004-06-30; First posted 2004-07-02 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Liver Transplantation
Keywords: Liver; Transplant
MeSH Terms: interventions — Sirolimus; Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Sirolimus (Rapamune)
- B (Active Comparator)
  Interventions: Drug: Cyclosporine or Tacrolimus

INTERVENTIONS:
Drug: Sirolimus (Rapamune)
  Arms: A
Drug: Cyclosporine or Tacrolimus
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the sirolimus conversion regimen as compared with the calcineurin inhibitor continuation regimen with regards to renal function in stable liver transplant subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 13 years (age greater than 18 years as required by some local regulations).
* Receiving immunosuppressive therapy with calcineurin inhibitors (CI) +/- corticosteroids +/- antimetabolite.
* 6 to 144 months after orthotopic liver transplantation.
* Cockcroft-Gault GFR values ≥40 mL/min and ≤90mL/min at screening

Exclusion Criteria:

* History of nonhepatic transplantation
* Evidence of systemic infection (sepsis, bacteremia, pneumonia etc).
* Known or suspected malignancy < 5 years before random assignment.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2002-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Italy, decresg@wyeth.com; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Czech Republic, WPPGCLI@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com
Locations (40):
- United States (10):
  - San Francisco, California
  - Tampa, Florida
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Rochester, Minnesota
  - Omaha, Nebraska
  - New York, New York
  - Rochester, New York
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
- Ghent, Belgium
- Canada (3):
  - Edmonton, Alberta
  - London, Ontario
  - Toronto, Ontario
- Prague, Czechia
- France (6):
  - Clichy
  - Lyon
  - Nice
  - Paris
  - Rennes
  - Villejuif
- Germany (3):
  - Berlin
  - Hamburg
  - München
- Italy (3):
  - Bologna
  - Milan
  - Padua
- Leiden, Netherlands
- Portugal (2):
  - Coimbra
  - Lisbon
- Spain (5):
  - Barcelona
  - Madrid
  - Pamplona
  - Santiago de Compostela
  - Valencia
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (3):
  - Birmingham
  - Edinburgh
  - Leeds

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited October 2002 to November 2006.
Pre-assignment Details: Patients were screened up to 30 days.
Groups:
- Sirolimus (SRL) Conversion: Sirolimus was administered once daily. A loading dose of sirolimus, 10 to 15 mg, was administered in divided doses on day 1: the first dose was given after collection of the sirolimus trough level and a minimum of 4 hours following the last dose of CNI, and the second dose approximately 12 hours after the first dose. On days 2 through 6, sirolimus was administered in a dose of 3 to 5 mg/day. For the remaining study period, day 7 through month 72, appropriate daily doses of sirolimus were administered to attain the recommended trough concentrations of 8 to 16 ng/mL (using a chromatographic method) or 10 to 20 ng/mL (using an immunoassay).
- Calcineurin Inhibitors (CNI) Continuation: Calcineurin Inhibitors administered per local practice to attain target trough levels of 3 to 10 ng/mL (tacrolimus) or 50 to 250 ng/mL (cyclosporin A), respectively.
Period: Randomization
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Started | 393 | 214
Completed | 389 | 210
Not Completed | 4 | 4
Not completed — Did not receive test article | 4 | 4
Period: Patients Dosed With Test Article
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Started | 389 | 210
Completed | 249 | 187
Not Completed | 140 | 23
Not completed — Adverse Event | 94 | 11
Not completed — Lost to Follow-up | 1 | 3
Not completed — Nonmedical event | 7 | 3
Not completed — Withdrawal by Subject | 16 | 3
Not completed — Protocol Violation | 11 | 3
Not completed — Lack of Efficacy | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation | Total
Number analyzed (Participants) | 393 | 214 | 607
Age Continuous [Median (Full Range); unit: years] | 57.0 [23.0 to 76.0] | 56.5 [21.0 to 73.0] | 57.0 [21.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 64 | 186.0
  Male | 271 | 150 | 421.0
Mean serum creatinine levels [Mean (Standard Deviation); unit: μmol/L] | 122.9 (32.3) | 125.2 (31.9) | 123.7 (32.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Adjusted Mean in Glomerular Filtration Rate (GFR)
Description: GFR is an index of kidney function. GFR was calculated using Cockcroft-Gault method. A normal GFR is >90 mL/min, higher values indicate better function. Change=adjusted mean of 12 months minus baseline. Mean adjusted for baseline GFR, with antimetabolite therapy status and hepatitis C status as fixed effects.
Time Frame: Baseline and 12 months
Population: The intent to treat population was analyzed and consisted of all patients randomly assigned to treatment. Patients were stratified by hepatitis C status and whether or not they were receiving antimetabolite therapy at time of randomization.
Measure: Mean (Standard Error); unit: mL/min
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Number analyzed (Participants) | 393 | 214
mL/min | -4.45 (1.12) | -3.07 (1.36)
Statistical Analysis 1: Comparison: Sirolimus (SRL) Conversion vs Calcineurin Inhibitors (CNI) Continuation; Test type: Superiority or Other; p = 0.342, Rank ANCOVA

2. Secondary Outcome: Number of Patients With a Biopsy Confirmed Acute Rejection
Description: Overall event rate is determined as yes or no.
Time Frame: 12 months
Population: The analysis population is the intent to treat. Any patient whose clinical rejection data was incomplete was designated as an acute rejection in the analysis.
Measure: Number; unit: patients
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Number analyzed (Participants) | 393 | 214
patients
  Yes | 46 | 13
  No | 347 | 201
Statistical Analysis 1: Comparison: Sirolimus (SRL) Conversion vs Calcineurin Inhibitors (CNI) Continuation; Comparison between treatment groups of percentages of patients with biopsy-confirmed acute rejection; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel

3. Secondary Outcome: Mean Serum Creatinine
Description: Observed mean values for serum creatinine.
Time Frame: 12 months
Population: On-therapy population; consisted of patients who were still receiving study medication at the defined endpoint.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Number analyzed (Participants) | 262 | 190
µmol/L | 119.0 (38.9) | 122.4 (31.5)
Statistical Analysis 1: Comparison: Sirolimus (SRL) Conversion vs Calcineurin Inhibitors (CNI) Continuation; Test type: Superiority or Other; p > 0.05, 1 way ANOVA, two sided

4. Primary Outcome: Patient and Graft Survival
Description: Endpoint was a composite assessment of patient and graft survival. Patients categorized as graft survival or graft loss. Graft loss defined as pure graft loss (requiring retransplant) or death (with a functioning graft), if the event occurred in the first 12 months after randomization. Patients with missing graft data were counted as graft losses.
Time Frame: 12 months
Population: Intent to treat analysis population with stratification by antimetabolite therapy and hepatitis C status.
Measure: Number; unit: patients
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Number analyzed (Participants) | 393 | 214
patients
  Graft survival | 367 | 202
  Graft loss (total) | 26 | 12
  Graft loss: Pure (with retransplant) | 0 | 0
  Graft loss: Death | 13 | 3
  Graft loss: Incomplete data | 13 | 9
Statistical Analysis 1: Comparison: Sirolimus (SRL) Conversion vs Calcineurin Inhibitors (CNI) Continuation; Test type: Non-Inferiority or Equivalence — The a priori criterion for declaring non-inferiority was a lower bound of the 95% confidence interval (CI) having a ≥ 5% difference in graft loss. -5.2 is < 5 % difference; Mean Difference (Net) = -1.2, 95% CI [-5.2 to 2.8] — Weighted difference in percentage of graft loss: (CNI% minus SRL%); negative values are favorable to CNI group

ADVERSE EVENTS:
Arm/Group | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Serious Adverse Events (participants affected / at risk) | 193 | 79
Other Adverse Events (participants affected / at risk) | 386/389 | 201/210
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sirolimus (SRL) Conversion | Calcineurin Inhibitors (CNI) Continuation
Abdominal pain (General disorders) | 10/389 | 4/210
Abdominal syndrome acute (General disorders) | 1/389 | 1/210
Abscess (General disorders) | 5/389 | 0/210
Accidental injury (General disorders) | 6/389 | 3/210
Accidental overdose (General disorders) | 3/389 | 0/210
Adenoma (General disorders) | 1/389 | 0/210
Allergic reaction (General disorders) | 1/389 | 0/210
Ascites (General disorders) | 1/389 | 0/210
Asthenia (General disorders) | 2/389 | 2/210
Back pain (General disorders) | 3/389 | 0/210
Carcinoma (General disorders) | 2/389 | 0/210
Cellulitis (General disorders) | 6/389 | 3/210
Chest pain (General disorders) | 4/389 | 3/210
Chills (General disorders) | 2/389 | 3/210
Death (General disorders) | 1/389 | 0/210
Diarrhea infectious (General disorders) | 1/389 | 0/210
Face edema (General disorders) | 1/389 | 0/210
Fever (General disorders) | 16/389 | 8/210
Flu syndrome (General disorders) | 1/389 | 0/210
Headache (General disorders) | 2/389 | 0/210
Hernia (General disorders) | 11/389 | 3/210
Infection (General disorders) | 10/389 | 2/210
Medication error (General disorders) | 1/389 | 0/210
Neck pain (General disorders) | 1/389 | 0/210
Neoplasm (General disorders) | 3/389 | 0/210
Overdose (General disorders) | 3/389 | 0/210
Pain (General disorders) | 4/389 | 0/210
Sepsis (General disorders) | 9/389 | 3/210
Septic shock (General disorders) | 1/389 | 0/210
Transplant rejection (General disorders) | 1/389 | 1/210
Angina pectoris (Cardiac disorders) | 3/389 | 1/210
Aortic stenosis (Vascular disorders) | 1/389 | 0/210
Arterial anomaly (Cardiac disorders) | 1/389 | 1/210
Arterial thrombosis (Vascular disorders) | 2/389 | 0/210
Atrial fibrillation (Cardiac disorders) | 1/389 | 1/210
Atrial flutter (Cardiac disorders) | 1/389 | 0/210
AV block (Cardiac disorders) | 1/389 | 0/210
AV block complete (Cardiac disorders) | 1/389 | 1/210
Cardiomegaly (Cardiac disorders) | 0/389 | 1/210
Cardiomyopathy (Cardiac disorders) | 1/389 | 0/210
Cardiovascular disorder (Cardiac disorders) | 3/389 | 0/210
Cerebral ischemia (Cardiac disorders) | 0/389 | 1/210
Cerebrovascular accident (Vascular disorders) | 1/389 | 6/210
Coronary occlusion (Cardiac disorders) | 1/389 | 1/210
Deep vein thrombosis (Vascular disorders) | 0/389 | 1/210
Heart failure (Cardiac disorders) | 4/389 | 1/210
Hemorrhage (Vascular disorders) | 3/389 | 1/210
Hypertension (Vascular disorders) | 2/389 | 1/210
Hypotension (Vascular disorders) | 1/389 | 0/210
Left heart failure (Cardiac disorders) | 1/389 | 0/210
Mesenteric venous occlusion (Vascular disorders) | 1/389 | 0/210
Myocardial infarct (Cardiac disorders) | 0/389 | 1/210
Myocardial ischemia (Cardiac disorders) | 2/389 | 0/210
Pericardial effusion (Cardiac disorders) | 1/389 | 0/210
Pericarditis (Cardiac disorders) | 1/389 | 1/210
Peripheral vascular disorder (Vascular disorders) | 1/389 | 0/210
Postural hypotension (Vascular disorders) | 1/389 | 0/210
Pulmonary embolus (Vascular disorders) | 0/389 | 2/210
Pulmonary hypertension (Vascular disorders) | 1/389 | 0/210
Shock (Cardiac disorders) | 1/389 | 0/210
Sick sinus syndrome (Cardiac disorders) | 1/389 | 0/210
Supraventricular tachycardia (Cardiac disorders) | 0/389 | 1/210
Syncope (Cardiac disorders) | 3/389 | 1/210
Tachycardia (Cardiac disorders) | 0/389 | 1/210
Vascular disorder (Vascular disorders) | 0/389 | 1/210
Carcinoma of the mouth (Gastrointestinal disorders) | 0/389 | 1/210
Cholangitis (Gastrointestinal disorders) | 5/389 | 2/210
Cholelithiasis (Gastrointestinal disorders) | 2/389 | 0/210
Colitis (Gastrointestinal disorders) | 2/389 | 1/210
Constipation (Gastrointestinal disorders) | 1/389 | 0/210
Diarrhea (Gastrointestinal disorders) | 16/389 | 5/210
Enteritis (Gastrointestinal disorders) | 0/389 | 1/210
Esophageal stenosis (Gastrointestinal disorders) | 1/389 | 0/210
Gamma glutamyl transpeptidase increased (Gastrointestinal disorders) | 3/389 | 0/210
Gastroenteritis (Gastrointestinal disorders) | 9/389 | 4/210
Gastrointestinal carcinoma (Gastrointestinal disorders) | 4/389 | 4/210
Gastrointestinal disorder (Gastrointestinal disorders) | 8/389 | 1/210
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 4/389 | 2/210
Hepatic neoplasia (Gastrointestinal disorders) | 3/389 | 2/210
Hepatitis (Gastrointestinal disorders) | 2/389 | 1/210
Ileitis (Gastrointestinal disorders) | 0/389 | 1/210
Ileus (Gastrointestinal disorders) | 3/389 | 1/210
Intestinal obstruction (Gastrointestinal disorders) | 2/389 | 1/210
Jaundice (Gastrointestinal disorders) | 0/389 | 1/210
Liver damage (Gastrointestinal disorders) | 1/389 | 1/210
Liver fatty deposit (Gastrointestinal disorders) | 1/389 | 0/210
Liver function tests abnormal (Gastrointestinal disorders) | 15/389 | 3/210
Melena (Gastrointestinal disorders) | 0/389 | 1/210
Nausea (Gastrointestinal disorders) | 6/389 | 1/210
Nausea and vomiting (Gastrointestinal disorders) | 0/389 | 1/210
Pancreatitis (Gastrointestinal disorders) | 2/389 | 0/210
Peridontal abcess (Gastrointestinal disorders) | 1/389 | 0/210
Rectal disorder (Gastrointestinal disorders) | 1/389 | 2/210
Diabetes mellitus (Endocrine disorders) | 3/389 | 2/210
Thyroid disorder (Endocrine disorders) | 0/389 | 1/210
Anemia (Blood and lymphatic system disorders) | 12/389 | 4/210
Aplastic anema (Blood and lymphatic system disorders) | 0/389 | 1/210
Coagulation disorder (Blood and lymphatic system disorders) | 0/389 | 1/210
International normalized ratio increased (Blood and lymphatic system disorders) | 1/389 | 0/210
Leukopenia (Blood and lymphatic system disorders) | 1/389 | 0/210
Lymphadenopathy (Blood and lymphatic system disorders) | 2/389 | 0/210
Lymphagitis (Blood and lymphatic system disorders) | 1/389 | 0/210
Microcytic anemia (Blood and lymphatic system disorders) | 1/389 | 0/210
Pancytopenia (Blood and lymphatic system disorders) | 1/389 | 1/210
Acidosis (Metabolism and nutrition disorders) | 1/389 | 0/210
Alkaline phosphotase increased (Metabolism and nutrition disorders) | 7/389 | 0/210
Bilirubinemia (Metabolism and nutrition disorders) | 0/389 | 1/210
BUN increased (Metabolism and nutrition disorders) | 2/389 | 0/210
Creatinine increased (Metabolism and nutrition disorders) | 5/389 | 2/210
Dehydration (Metabolism and nutrition disorders) | 4/389 | 3/210
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/389 | 0/210
Electrolyte abnormality (Metabolism and nutrition disorders) | 1/389 | 0/210
Gout (Metabolism and nutrition disorders) | 0/389 | 1/210
Healing abnormal (Metabolism and nutrition disorders) | 5/389 | 2/210
Hyperglycemia (Metabolism and nutrition disorders) | 2/389 | 1/210
Hyperkalemia (Metabolism and nutrition disorders) | 0/389 | 1/210
Hyperlipemia (Metabolism and nutrition disorders) | 1/389 | 0/210
Hypocalcemia (Metabolism and nutrition disorders) | 1/389 | 0/210
Hypoglycemia (Metabolism and nutrition disorders) | 2/389 | 0/210
Hypokalemia (Metabolism and nutrition disorders) | 3/389 | 0/210
Hyponatremia (Metabolism and nutrition disorders) | 0/389 | 1/210
Peripheral edema (Metabolism and nutrition disorders) | 4/389 | 0/210
SGOT increased (Metabolism and nutrition disorders) | 6/389 | 2/210
SGPT increased (Metabolism and nutrition disorders) | 5/389 | 2/210
Weight gain (Metabolism and nutrition disorders) | 0/389 | 1/210
Weight loss (Metabolism and nutrition disorders) | 1/389 | 1/210
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/389 | 2/210
Arthritis (Musculoskeletal and connective tissue disorders) | 2/389 | 0/210
Arthrosis (Musculoskeletal and connective tissue disorders) | 2/389 | 2/210
Bone necrosis (Musculoskeletal and connective tissue disorders) | 1/389 | 0/210
Bursitis (Musculoskeletal and connective tissue disorders) | 1/389 | 0/210
Musculoskeletal anomaly (Musculoskeletal and connective tissue disorders) | 1/389 | 0/210
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0/389 | 1/210
Alcoholism (Nervous system disorders) | 1/389 | 0/210
Aphasia (Nervous system disorders) | 0/389 | 1/210
CNS neoplasia (Nervous system disorders) | 0/389 | 1/210
Convulsion (Nervous system disorders) | 2/389 | 1/210
Depression (Nervous system disorders) | 1/389 | 1/210
Dizziness (Nervous system disorders) | 1/389 | 1/210
Dysarthria (Nervous system disorders) | 0/389 | 1/210
Hemiplegia (Nervous system disorders) | 0/389 | 1/210
Hypesthesia (Nervous system disorders) | 1/389 | 0/210
Subdural hematoma (Nervous system disorders) | 1/389 | 0/210
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0/389 | 2/210
Carcinoma of lung (Respiratory, thoracic and mediastinal disorders) | 3/389 | 2/210
Cough increased (Respiratory, thoracic and mediastinal disorders) | 3/389 | 1/210
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7/389 | 1/210
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/389 | 1/210
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2/389 | 0/210
Lung edema (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Lung hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Lung infiltration nos (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2/389 | 0/210
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2/389 | 0/210
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 17/389 | 4/210
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2/389 | 0/210
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1/389 | 0/210
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5/389 | 1/210
Herpes simplex (Skin and subcutaneous tissue disorders) | 1/389 | 0/210
Herpes zoster (Skin and subcutaneous tissue disorders) | 1/389 | 1/210
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1/389 | 0/210
Purpuric rash (Skin and subcutaneous tissue disorders) | 0/389 | 1/210
Rash (Skin and subcutaneous tissue disorders) | 3/389 | 1/210
Skin carcinoma (Skin and subcutaneous tissue disorders) | 14/389 | 19/210
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1/389 | 0/210
Skin melanoma (Skin and subcutaneous tissue disorders) | 1/389 | 3/210
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/389 | 0/210
Cataract specified (Eye disorders) | 1/389 | 1/210
Eye hemorrhage (Eye disorders) | 1/389 | 0/210
Glaucoma (Eye disorders) | 1/389 | 0/210
Retinal detachment (Eye disorders) | 1/389 | 0/210
Retinal disorder (Eye disorders) | 1/389 | 0/210
Acute kidney failure (Renal and urinary disorders) | 7/389 | 2/210
Albuminuria (Renal and urinary disorders) | 1/389 | 0/210
Breast neoplasm (Reproductive system and breast disorders) | 0/389 | 1/210
Dysuria (Renal and urinary disorders) | 1/389 | 1/210
Fallopian tube disorder (Reproductive system and breast disorders) | 1/389 | 0/210
Hematuria (Renal and urinary disorders) | 0/389 | 1/210
Hydronephrosis (Renal and urinary disorders) | 1/389 | 1/210
Kidney calculus (Renal and urinary disorders) | 3/389 | 1/210
Kidney failure (Renal and urinary disorders) | 7/389 | 1/210
Kidney function abnormal (Renal and urinary disorders) | 6/389 | 1/210
Nephritis (Renal and urinary disorders) | 1/389 | 0/210
Nephrosclerosis (Renal and urinary disorders) | 2/389 | 0/210
Nephrosis (Renal and urinary disorders) | 1/389 | 0/210
Ovarian cyst (Reproductive system and breast disorders) | 3/389 | 0/210
Ovarian disorder (Reproductive system and breast disorders) | 0/389 | 1/210
Polyuria (Renal and urinary disorders) | 1/389 | 0/210
Prostatic carcinoma (Reproductive system and breast disorders) | 3/389 | 0/210
Prostatic disorder (Reproductive system and breast disorders) | 0/389 | 1/210
Pyelonephritis (Renal and urinary disorders) | 1/389 | 0/210
Unintended pregnancy (Reproductive system and breast disorders) | 0/389 | 1/210
Uremia (Renal and urinary disorders) | 2/389 | 1/210
Urinary tract disorder (Renal and urinary disorders) | 0/389 | 1/210
Urinary tract infection (Renal and urinary disorders) | 7/389 | 3/210
Urine abnormality (Renal and urinary disorders) | 1/389 | 0/210
Urolithiasis (Renal and urinary disorders) | 1/389 | 0/210
Device malfunction (General disorders) | 1/389 | 1/210
Local reaction to procedure (General disorders) | 13/389 | 3/210
Surgical procedure (General disorders) | 1/389 | 0/210
Rectal hemorrhage (Gastrointestinal disorders) | 0/389 | 1/210
Sclerosing cholangitis (Gastrointestinal disorders) | 1/389 | 0/210
Stomatitis (Gastrointestinal disorders) | 1/389 | 0/210
Stools abnormal (Gastrointestinal disorders) | 1/389 | 0/210
Ulcerative colitis (Gastrointestinal disorders) | 1/389 | 2/210
Vomiting (Gastrointestinal disorders) | 10/389 | 2/210
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus (SRL) Conversion (N=389) | Calcineurin Inhibitors (CNI) Continuation (N=210)
Abdominal pain (General disorders) | 70 | 30
Accidental injury (General disorders) | 67 | 32
Asthenia (General disorders) | 79 | 28
Back pain (General disorders) | 42 | 27
Chest pain (General disorders) | 31 | 18
Face edema (General disorders) | 22 | 4
Fever (General disorders) | 79 | 26
Flu syndrome (General disorders) | 22 | 7
Headache (General disorders) | 84 | 23
Hernia (General disorders) | 25 | 10
Pain (General disorders) | 71 | 39
Hypertension (Cardiac disorders) | 65 | 40
Anorexia (Gastrointestinal disorders) | 25 | 5
Aphthous stomatitis (Gastrointestinal disorders) | 34 | 2
Constipation (Gastrointestinal disorders) | 36 | 20
Diarrhea (Gastrointestinal disorders) | 136 | 38
Dyspepsia (Gastrointestinal disorders) | 17 | 11
Gastrointestinal disorder (Gastrointestinal disorders) | 26 | 10
Liver function tests abnormal (Gastrointestinal disorders) | 59 | 25
Mouth ulceration (Gastrointestinal disorders) | 44 | 2
Nausea (Gastrointestinal disorders) | 51 | 19
Stomatitis (Gastrointestinal disorders) | 103 | 4
Vomiting (Gastrointestinal disorders) | 35 | 17
Diabetes mellitus (Endocrine disorders) | 25 | 9
Anemia (Blood and lymphatic system disorders) | 94 | 19
Leukopenia (Blood and lymphatic system disorders) | 55 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 58 | 8
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 32 | 10
BUN increased (Metabolism and nutrition disorders) | 12 | 13
Creatinine increased (Metabolism and nutrition disorders) | 24 | 26
Hypercholesteremia (Metabolism and nutrition disorders) | 110 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 39 | 22
Hyperkalemia (Metabolism and nutrition disorders) | 11 | 17
Hyperlipemia (Metabolism and nutrition disorders) | 159 | 20
Hyperuricemia (Metabolism and nutrition disorders) | 10 | 16
Hypokalemia (Metabolism and nutrition disorders) | 23 | 5
Lactic dehydrogenase increased (Metabolism and nutrition disorders) | 20 | 3
Peripheral edema (Metabolism and nutrition disorders) | 127 | 29
SGOT increased (Metabolism and nutrition disorders) | 37 | 12
SGPT increased (Metabolism and nutrition disorders) | 40 | 9
Weight loss (Metabolism and nutrition disorders) | 26 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 35
Leg cramps (Musculoskeletal and connective tissue disorders) | 5 | 12
Depression (Nervous system disorders) | 16 | 13
Dizziness (Nervous system disorders) | 36 | 15
Insomnia (Nervous system disorders) | 27 | 11
Paresthesia (Nervous system disorders) | 20 | 4
Cough increased (Respiratory, thoracic and mediastinal disorders) | 66 | 28
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 36 | 13
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 40 | 14
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 35 | 11
Acne (Skin and subcutaneous tissue disorders) | 52 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 3
Erythema (Respiratory, thoracic and mediastinal disorders) | 24 | 3
Pruritus (Respiratory, thoracic and mediastinal disorders) | 50 | 14
Rash (Skin and subcutaneous tissue disorders) | 111 | 16
Skin disorder (Skin and subcutaneous tissue disorders) | 28 | 13
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 8 | 12
Albuminuria (Renal and urinary disorders) | 25 | 5
Kidney function abnormal (Renal and urinary disorders) | 24 | 22
Local reaction to procedure (Injury, poisoning and procedural complications) | 36 | 16
Cellulitis (General disorders) | 20 | 7
Flu Syndrome (General disorders) | 16 | 15
Infection (General disorders) | 97 | 43
Gastroenteritis (Gastrointestinal disorders) | 19 | 12
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 25 | 14
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 30 | 9
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 27 | 15
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 54 | 36
Herpes Simplex (Skin and subcutaneous tissue disorders) | 33 | 3
Urinary Tract Infection (Renal and urinary disorders) | 36 | 21
Skin Carcinoma (Skin and subcutaneous tissue disorders) | 14 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.